CLINICAL TRIAL: NCT04070820
Title: "Combination Treatment for Enterococcus Faecalis Bacteremia: a Prospective, Multicenter, Observational Study"
Brief Title: Combination Treatment for Enterococcus Faecalis Bacteriemia Multicenter, Observational Study"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Michele Bartoletti, Assistant Professor, University of Bologna
Other Study IDs: EfFAECT
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Enterococcal Bacteraemia; Enterococcus Faecalis Infection; Enterococcal Endocarditis; Bloodstream Infection
Keywords: Combination therapy; Bloodstream Infection; Enterococcus faecalis Infection; Endocarditis
MeSH Terms: conditions — Sepsis; Endocarditis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, multicenter, observational study on the evaluation of efficacy of appropriate monotherapy vs combination treatment for non-complicated Enterococcus faecalis bloodstream infection (EF-BSI).

The aims of our study are:

Primary:

To compare the efficacy of appropriate monotherapy vs combination treatment for EF-BSI, according to standard of care.

Secondary:

1. To compare the impact on clinical outcome of the initial combination therapy in the subgroup of patients with enterococcal endocarditis. In this case we will evaluate only the antibiotic treatment administered before the diagnosis of endocarditis assuming that any case of endocarditis will be treated with a combination therapy.
2. To compare the efficacy of combination treatment (vs monotherapy) in the following subgroup of patients:

   A. Patients with low versus high risk of endocarditis according with the "Number of positive blood cultures, Origin of the bacteremia, previous Valve disease, Auscultation of heart murmur (NOVA) score".

   B. Patients with metastatic septic localizations. C. Patients with catheter-related BSI. D. Patients with indwelling cardiovascular device or prosthetic valve.
3. To validate the NOVA score as a predictor of enterococcal endocarditis in a large multicentre cohort of patients with EF-BSI.
4. To estimate optimal duration of treatment of EF-BSI in patients without endocarditis.
5. To evaluate the rate of 90-day development of Clostridium difficile infection.

The promoting center is S. Orsola-Malpighi Hospital is a 1,420-bed tertiary care University Hospital in Bologna with an average of 72,000 admissions per year. A dedicate team of Infectious Diseases (ID) specialists is active in the promoting center. Investigators of this team have already coordinated multicenter studies on infections topics. Centers from other countries will be invited to participate by email, they will be ask to fulfil an agreement form.

All consecutive, unselected patients with monomicrobial EF-BSI will be screened for study inclusion. We expect to enroll about 500 patients.

Period of data collection will be from september 2019 to 31th December 2020.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years)
* First monomicrobial EF-BSI
* Receipt of ≥ 5 days of at least one in vitro active drug (ampicillin, amoxicillin/clavulanate, ampicillin/sulbactam, piperacillin, vancomycin, teicoplanin, daptomycin and linezolid) with or without a synergistic drug (ceftriaxone, gentamycin, streptomycin), at common suggested dosages for EF-BSI in empirical or definitive therapy
* Written informed consent

Exclusion Criteria:

* Short term (within 3 days from BSI) mortality
* Other concomitant infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive, unselected patients with a first episode of monomicrobial EF-BSI will be screened for study inclusion
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Survival | End of Treatment, at least 2 weeks from first negative follow-up bloodculture
  Patient alive
Body temperature (Celsius degrees) | End of Treatment, at least 2 weeks from first negative follow-up bloodculture
  Fever resolution
Sequential Organ Failure Assessment (SOFA) Score | End of Treatment, at least 2 weeks from first negative follow-up bloodculture
  Stable or improved SOFA score. Total SOFA score ranges from 0 to 24 points. Total SOFA score consist of the sum of individual score of following items: Respiratory System (PaO2/FiO2), Cardiovascular system (Mean Arterial Pressure or administration vasopressure required), Newrvous System (Glasgow Coma Scale), Liver (bilirubin), Coagulation (platelets), Kidneys (creatinine). Each items receive a score ranging from 0 to 4 pt.
Blood cultures | End of Treatment, at least 2 weeks from first negative follow-up bloodculture
  Follow-up Blood cultures negative for E. faecalis
Blood cultures | 90 days from End of Treatment
  No relapse of EF-BSI
Antibiotic therapy | 90 days from End of Treatment
  No need to modify initial therapy

CONTACTS AND LOCATIONS:
Overall Officials: Michele Bartoletti, Principal Investigator — Dipartimento di Scienze mediche e chirurgiche, Alma Mater-University of Bologna
Locations (1):
- Infectious Disease Unit - S.Orsola Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wisplinghoff H, Bischoff T, Tallent SM, Seifert H, Wenzel RP, Edmond MB. Nosocomial bloodstream infections in US hospitals: analysis of 24,179 cases from a prospective nationwide surveillance study. Clin Infect Dis. 2004 Aug 1;39(3):309-17. doi: 10.1086/421946. Epub 2004 Jul 15. PMID 15306996
- [Background] Rodriguez-Bano J, Lopez-Prieto MD, Portillo MM, Retamar P, Natera C, Nuno E, Herrero M, del Arco A, Munoz A, Tellez F, Torres-Tortosa M, Martin-Aspas A, Arroyo A, Ruiz A, Moya R, Corzo JE, Leon L, Perez-Lopez JA; SAEI/SAMPAC Bacteraemia Group. Epidemiology and clinical features of community-acquired, healthcare-associated and nosocomial bloodstream infections in tertiary-care and community hospitals. Clin Microbiol Infect. 2010 Sep;16(9):1408-13. doi: 10.1111/j.1469-0691.2009.03089.x. PMID 19845694
- [Background] Cahill TJ, Prendergast BD. Infective endocarditis. Lancet. 2016 Feb 27;387(10021):882-93. doi: 10.1016/S0140-6736(15)00067-7. Epub 2015 Sep 1. PMID 26341945
- [Background] Reigadas E, Rodriguez-Creixems M, Guembe M, Sanchez-Carrillo C, Martin-Rabadan P, Bouza E. Catheter-related bloodstream infection caused by Enterococcus spp. Clin Microbiol Infect. 2013 May;19(5):457-61. doi: 10.1111/j.1469-0691.2012.03897.x. Epub 2012 May 22. PMID 22612464
- [Background] Chirouze C, Athan E, Alla F, Chu VH, Ralph Corey G, Selton-Suty C, Erpelding ML, Miro JM, Olaison L, Hoen B; International Collaboration on Endocarditis Study Group. Enterococcal endocarditis in the beginning of the 21st century: analysis from the International Collaboration on Endocarditis-Prospective Cohort Study. Clin Microbiol Infect. 2013 Dec;19(12):1140-7. doi: 10.1111/1469-0691.12166. Epub 2013 Mar 20. PMID 23517406
- [Background] McBride SJ, Upton A, Roberts SA. Clinical characteristics and outcomes of patients with vancomycin-susceptible Enterococcus faecalis and Enterococcus faecium bacteraemia--a five-year retrospective review. Eur J Clin Microbiol Infect Dis. 2010 Jan;29(1):107-14. doi: 10.1007/s10096-009-0830-5. Epub 2009 Nov 15. PMID 19916034
- [Background] Gray J, Marsh PJ, Stewart D, Pedler SJ. Enterococcal bacteraemia: a prospective study of 125 episodes. J Hosp Infect. 1994 Jul;27(3):179-86. doi: 10.1016/0195-6701(94)90125-2. PMID 7963458
- [Background] Suppli M, Aabenhus R, Harboe ZB, Andersen LP, Tvede M, Jensen JU. Mortality in enterococcal bloodstream infections increases with inappropriate antimicrobial therapy. Clin Microbiol Infect. 2011 Jul;17(7):1078-83. doi: 10.1111/j.1469-0691.2010.03394.x. Epub 2010 Dec 3. PMID 20946408
- [Background] Foo H, Chater M, Maley M, van Hal SJ. Glycopeptide use is associated with increased mortality in Enterococcus faecalis bacteraemia--authors' response. J Antimicrob Chemother. 2014 Nov;69(11):3166. doi: 10.1093/jac/dku329. Epub 2014 Aug 12. No abstract available. PMID 25118271
- [Background] Cheah AL, Spelman T, Liew D, Peel T, Howden BP, Spelman D, Grayson ML, Nation RL, Kong DC. Enterococcal bacteraemia: factors influencing mortality, length of stay and costs of hospitalization. Clin Microbiol Infect. 2013 Apr;19(4):E181-9. doi: 10.1111/1469-0691.12132. Epub 2013 Feb 7. PMID 23398607
- [Background] Mermel LA, Allon M, Bouza E, Craven DE, Flynn P, O'Grady NP, Raad II, Rijnders BJ, Sherertz RJ, Warren DK. Clinical practice guidelines for the diagnosis and management of intravascular catheter-related infection: 2009 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jul 1;49(1):1-45. doi: 10.1086/599376. PMID 19489710
- [Background] Murray BE. The life and times of the Enterococcus. Clin Microbiol Rev. 1990 Jan;3(1):46-65. doi: 10.1128/CMR.3.1.46. PMID 2404568
- [Background] Gavalda J, Len O, Miro JM, Munoz P, Montejo M, Alarcon A, de la Torre-Cisneros J, Pena C, Martinez-Lacasa X, Sarria C, Bou G, Aguado JM, Navas E, Romeu J, Marco F, Torres C, Tornos P, Planes A, Falco V, Almirante B, Pahissa A. Brief communication: treatment of Enterococcus faecalis endocarditis with ampicillin plus ceftriaxone. Ann Intern Med. 2007 Apr 17;146(8):574-9. doi: 10.7326/0003-4819-146-8-200704170-00008. PMID 17438316
- [Background] Maki DG, Agger WA. Enterococcal bacteremia: clinical features, the risk of endocarditis, and management. Medicine (Baltimore). 1988 Jul;67(4):248-69. PMID 3134590
- [Background] Sandoe JA, Witherden IR, Au-Yeung HK, Kite P, Kerr KG, Wilcox MH. Enterococcal intravascular catheter-related bloodstream infection: management and outcome of 61 consecutive cases. J Antimicrob Chemother. 2002 Oct;50(4):577-82. doi: 10.1093/jac/dkf182. PMID 12356804
- [Background] Ibrahim SL, Zhang L, Brady TM, Hsu AJ, Cosgrove SE, Tamma PD. Low-dose Gentamicin for Uncomplicated Enterococcus faecalis Bacteremia May be Nephrotoxic in Children. Clin Infect Dis. 2015 Oct 1;61(7):1119-24. doi: 10.1093/cid/civ461. Epub 2015 Jun 16. PMID 26082503
- [Background] Diallo K, Kern WV, de With K, Luc A, Thilly N, Pulcini C; ESGAP and ESGBIS. Management of bloodstream infections by infection specialists in France and Germany: a cross-sectional survey. Infection. 2018 Jun;46(3):333-339. doi: 10.1007/s15010-018-1122-8. Epub 2018 Feb 3. PMID 29397537
- [Background] Diallo K, Thilly N, Luc A, Beraud G, Ergonul O, Giannella M, Kofteridis D, Kostyanev T, Pano-Pardo JR, Retamar P, Kern W, Pulcini C; ESGAP, ESGBIS. Management of bloodstream infections by infection specialists: an international ESCMID cross-sectional survey. Int J Antimicrob Agents. 2018 May;51(5):794-798. doi: 10.1016/j.ijantimicag.2017.12.010. Epub 2018 Jan 5. PMID 29309899
- [Background] Bouza E, Kestler M, Beca T, Mariscal G, Rodriguez-Creixems M, Bermejo J, Fernandez-Cruz A, Fernandez-Aviles F, Munoz P; Grupo de Apoyo al Manejo de la Endocarditis. The NOVA score: a proposal to reduce the need for transesophageal echocardiography in patients with enterococcal bacteremia. Clin Infect Dis. 2015 Feb 15;60(4):528-35. doi: 10.1093/cid/ciu872. Epub 2014 Nov 7. PMID 25381321
- [Background] Friedman ND, Kaye KS, Stout JE, McGarry SA, Trivette SL, Briggs JP, Lamm W, Clark C, MacFarquhar J, Walton AL, Reller LB, Sexton DJ. Health care--associated bloodstream infections in adults: a reason to change the accepted definition of community-acquired infections. Ann Intern Med. 2002 Nov 19;137(10):791-7. doi: 10.7326/0003-4819-137-10-200211190-00007. PMID 12435215
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338